CLINICAL TRIAL: NCT01186575
Title: Text Messaging to Improve Adherence to Post-Operative Clinic Appointments and Reduce Early Resumption of Sexual Intercourse After Adult Male Circumcision: A Randomized Controlled Trial
Brief Title: Text Messaging to Improve Adherence to Clinic Visits and Reduce Early Resumption of Sexual Intercourse After Male Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Illinois at Chicago (Other); Kenya Medical Research Institute (Other)
Responsible Party: Principal Investigator, Thomas Odeny, Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 38465-E/G
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome; Circumcision, Male; Patient Compliance; Cellular Phone
Keywords: HIV Infections; Acquired Immunodeficiency Syndrome; Circumcision, Male; Coitus; Patient Compliance; Cellular Phone
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Patient Compliance; Coitus | interventions — Spermine Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text Message (Experimental): Context-sensitive text messages are sent to men after undergoing circumcision
  Interventions: Other: Text Message
- Usual Care (No Intervention): Usual care after adult male circumcision (no text messages)

INTERVENTIONS:
Other: Text Message — Context-sensitive text messages are sent to men after undergoing circumcision
  Other Names: SMS, short message service, text messaging
  Arms: Text Message

SUMMARY:
Male circumcision (MC) reduces, by more than half, the risk of HIV-1 acquisition. WHO and UNAIDS recommend that "male circumcision should be recognized as an efficacious intervention for HIV prevention especially in countries and regions with heterosexual HIV epidemics and low male circumcision prevalence." As a result, programs have been introduced and scaled up for voluntary medical male circumcision. Kenya leads with the largest expansion of services.

Early resumption of sexual intercourse after MC may have deleterious effects, including higher rates of post-operative surgical complications, and higher HIV acquisition among females in couples that resume sexual activity before certified wound healing. In the context of rapid scale-up of MC, adherence to post-operative clinic appointments allows clinicians to assess wound healing and to deliver risk reduction counseling. Abstinence from sexual intercourse before complete wound healing would reduce the rate of post-operative adverse events and minimize the risk of HIV transmission from HIV-infected men to their uninfected female partners.

To the investigators knowledge, the effect of reminders delivered via text messaging to promote adherence to clinic visits and abstinence after MC has not been investigated. The investigators propose a randomized controlled trial in which men who will have undergone voluntary medical male circumcision at selected sites in Kisumu will be randomized to receive either the intervention (context-sensitive text messages after circumcision) or the control condition (usual care). This study seeks to determine (a) the effect of regular text messages sent to men after circumcision on attendance of the scheduled 7-day post-operative clinic visit versus usual care; (b) the proportion of men who resume sexual activity before 42 days post-procedure after receiving regular text messages versus usual care within the 42 days post-circumcision; and (c) to identify potential predictors of failure to attend the scheduled 7-day post-operative visit and early resumption of sexual intercourse.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18 years or older
* Have undergone circumcision on the day they are screened for the study
* Currently own a mobile phone with text-messaging capability, and
* Have the mobile phone in their possession at the time of enrollment
* Able and willing to respond to a questionnaire administered via a phone call

Exclusion Criteria:

* Prior participation in a study on male circumcision
* Currently participating in other ongoing research studies
* Any medical condition or situation exists such that study participation would not be in the man's best interest, as determined by the investigator

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Proportion of men failing to return for a post-operative clinic visit at 7 days. | 7 days
  This proportion will be determined by examining each participant's clinic records after their 7th post-operative day. Adherence to this clinic visit will be analyzed as a dichotomous variable.
Proportion of men who report resumption of sexual activity before 42 days post-circumcision. | 42 days
  This proportion will be determined by self-report using a brief questionnaire delivered via phone call. The analysis will be as a dichotomous variable, with participants considered as having either 'resumed' or 'not resumed.'

SECONDARY OUTCOMES:
Time to resumption of sex by study arm | 42 days
Correlates of failure to attend the scheduled 7-day post-operative visit | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Odeny, MBChB, MPH, Principal Investigator — University of Washington; R S McClelland, MD, MPH, Study Chair — University of Washington; Elizabeth A Bukusi, MBChB, MMed, MPH, PhD, Study Chair — Kenya Medical Research Institute; Jane Simoni, PhD, Study Chair — University of Washington; King K Holmes, MD, PhD, Study Chair — University of Washington; Robert C Bailey, PhD, MPH, Study Chair — University of Illinois at Chicago
Locations (1):
- Nyanza Reproductive Health Society, Kisumu, Nyanza, Kenya

REFERENCES:
- [Result] Odeny TA, Bailey RC, Bukusi EA, Simoni JM, Tapia KA, Yuhas K, Holmes KK, McClelland RS. Text messaging to improve attendance at post-operative clinic visits after adult male circumcision for HIV prevention: a randomized controlled trial. PLoS One. 2012;7(9):e43832. doi: 10.1371/journal.pone.0043832. Epub 2012 Sep 5. PMID 22957034
- [Result] Odeny TA, Bailey RC, Bukusi EA, Simoni JM, Tapia KA, Yuhas K, Holmes KK, McClelland RS. Effect of text messaging to deter early resumption of sexual activity after male circumcision for HIV prevention: a randomized controlled trial. J Acquir Immune Defic Syndr. 2014 Feb 1;65(2):e50-7. doi: 10.1097/QAI.0b013e3182a0a050. PMID 23846561